CLINICAL TRIAL: NCT06888947
Title: Influence of Collagen Cone on the Outcomes of Immediate Dental Implant Placement in Esthetic Zone
Acronym: dental implant
Status: Enrolling by invitation | Type: Observational
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Hala Fathy Abd El Fattah, principal investigator, Faculty of Dental Medicine for Girls
Other Study IDs: 1445 AH - 2023 AG; 1234 (Other Grant/Funding Number: azhar university)
Record Dates: First submitted 2025-01-07; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-01

CONDITIONS: Immediate Implant Placement; Evaluate Buccal Bone Plate Around Dental Implant
Keywords: immediate implant; collagen cone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 8 patient will receive immediate implant with collagen cone.: 8 patient will receive immediate implant with collagen cone.
  Interventions: Procedure: use immediate implant in socket with collagen cone
- Control group 8 patient will receive immediate implant.: Control group 8 patient will receive immediate implant.

INTERVENTIONS:
Procedure: use immediate implant in socket with collagen cone — use immediate implant in socket with collagen cone
  Groups: 8 patient will receive immediate implant with collagen cone.

SUMMARY:
Influence of Collagen Cone on the Outcomes of Immediate Dental Implant Placement in Esthetic zone

DETAILED DESCRIPTION:
The present study will be performed to assess effect of collagen cone for bone width and length around immediate implants in esthetics zone.

ELIGIBILITY:
Inclusion Criteria:

- 1-Patients were free from any systemic disease as evidenced by Burket's oral medicine health history questionnaire 2- Each patient required extraction of a non-restorable premolar or anterior tooth maxilla and requested implant restoration.

3-All patients should not have any known contraindication to oral surgery. 4-Male or female with age range 30 - 50 years.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patient with unrestorable tooth/teeth in esthetic zone seeking tooth/teeth replacement.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2026-08-05 (Estimated)

PRIMARY OUTCOMES:
1- Clinical examination | 9 months
  Probing depth around the dental implant using graduated plastic periodontal probe (Keratinized Mucosa, bleeding on probing and gingival tissue condition)

SECONDARY OUTCOMES:
CBCT | 9 months
  Improvement of esthetic outcome using collagen cone impacted in the socket with immediate implant by measure the improvement of bone width, length and density.

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Gawish, professor, Study Director — Al-Azhar University; lobna Abd-El Aziz, Lecturer, Study Director — Al-Azhar University
Locations (1):
- Hala Fathy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided